CLINICAL TRIAL: NCT04992923
Title: Prospective Cohort Study of Patients With Infective Endocarditis Admitted at Cardiology Institute of Pitié-Salpêtrière Hospital
Brief Title: Prospective Cohort Study of Patients With Infective Endocarditis at Pitié-Salpêtrière Hospital
Acronym: EIPSL
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200685
Record Dates: First submitted 2020-11-05; First posted 2021-08-05 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Infective Endocarditis
Keywords: Infective endocarditis, prospective,; prognosis, biomarker, embolism
MeSH Terms: conditions — Endocarditis; Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infective endocarditis (IE) is a severe condition associated with high mortality. Due to the relative low prevalence of IE, prospective data are lacking and current guidelines are mostly based on expert consensus with low level of evidence. IE is also associated with severe complications especially strokes that occur in about one third of the patients.

In order to improve the management and the prognosis of IE, clinical data from larges prospective cohort studies are needed.

DETAILED DESCRIPTION:
The study will take place at the Cardiology institute of the Pitié-Salpêtrière hospital. All patients referred to this tertiary care center for IE management will be included.

The characteristics of the patients (demographics, clinical, laboratory, and imaging data) at the time of IE diagnosis and during the follow-up will be collected. The patients will be followed up to 10 years after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed IE according to European Society of Cardiology criteria

Exclusion Criteria:

* Opposition of the patient to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients with IE admitted at Cardiology institute of the Pitié-Salpêtrière hospital
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2040-09 (Estimated); Study Completion 2041-03 (Estimated)

PRIMARY OUTCOMES:
All-cause in hospital mortality | up to 90 days
  All-cause mortality during the length of hospital stay

SECONDARY OUTCOMES:
All-cause mortality | an average of 10 years
  mortality at longest follow-up
symptomatic or asymptomatic systemic embolism | up to 90 days after inclusion
  symptomatic or asymptomatic systemic embolism confirmed by any type of imaging during initial hospitalization
Association between coagulation biomarkers (D-dimer, fibrin monomer, circulating anticoagulant, von Willebrandt factor (VWF) antigen level, von Willebrandt factor (VWF) activity) assessed at the inclusion and the presence of systemic embolism | inclusion
  Association between coagulation biomarkers (D-dimer, fibrin monomer, circulating anticoagulant, von Willebrandt factor (VWF) antigen level, von Willebrandt factor (VWF) activity) assessed at the inclusion and the presence of systemic embolism at the admission Initial Hospitalization
Association between coagulation biomarkers (D-dimer, fibrin monomer, circulating anticoagulant, von Willebrandt factor (VWF) antigen level, von Willebrandt factor (VWF) activity) assessed at the inclusion and the presence of systemic embolism | up to 90 days after inclusion
  Association between coagulation biomarkers(D-dimer, fibrin monomer, circulating anticoagulant, von Willebrandt factor (VWF) antigen level, von Willebrandt factor (VWF) activity) assessed at the inclusion and the presence of systemic embolism within 90 days after admission
heart failure, intracranial hemorrhage, or false vascular aneurysm during hospitalization | up to 90 days after inclusion
  Occurrence of heart failure, intracranial hemorrhage, or false vascular aneurysm during the length of hospital stay
Stroke | 90 days after inclusion
  Stroke during the length of hospital stay
composite criteria of stroke, Intracranial hemorrhage, hospitalization due to cardiovascular cause or IE recurrence | 1 year after inclusion
  Occurrence of a composite criteria of stroke, Intracranial hemorrhage, hospitalization due to cardiovascular cause or IE recurrence at one year
composite criteria of stroke, Intracranial hemorrhage, hospitalization due to cardiovascular cause or IE recurrence | through study completion, an average of 10 years
  Occurrence of a composite criteria of stroke, Intracranial hemorrhage, hospitalization due to cardiovascular cause or IE recurrence at the longest follow-up
composite criteria of all-cause mortality, stroke or intracranial hemorrhage, severe hemorrhage as defined by BARC score ≥ 3 | 1 year after inclusion
  on-year composite criteria of all-cause mortality, stroke or intracranial hemorrhage, severe hemorrhage as defined by BARC score ≥ 3
composite criteria of all-cause mortality, stroke or intracranial hemorrhage, severe hemorrhage as defined by BARC score ≥ 3 | through study completion, an average of 10 years
  Occurrence of a composite criteria of all-cause mortality, stroke or intracranial hemorrhage, severe hemorrhage as defined by BARC score ≥ 3 at the longest follow-up
Association between occurrence of systemic embolism and the composite criteria of all-cause mortality, stroke or intracranial hemorrhage, severe hemorrhage as defined by BARC score ≥ 3 | 1 year after inclusion
  Association between occurrence of systemic embolism and the composite criteria of all-cause mortality, stroke or intracranial hemorrhage, severe hemorrhage as defined by BARC score ≥ 3 at one year
Occurrence of contrast-associated acute kidney injury during the length of hospital stay | up to 90 days after inclusion
  rise of serum creatinine > 26.5 mcmol/L or > 50% elevation from baseline over the course of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Nadjib Hammoudi, MD, PhD, Principal Investigator — Pitié-Salpêtrière Hospital (AP-HP)
Locations (1):
- APHP Pitié-Salpêtrière Hospital, Department of Cardiology, Paris, France

IPD SHARING:
Plan to Share IPD: No